CLINICAL TRIAL: NCT02231177
Title: A Randomised, Double-blind, 3-way Crossover Study to Compare Pharmacokinetics and Safety of 10 μg BI 1744 CL Plus 5 μg Tiotropium Bromide Given as Fixed Dose Combination Via the Respimat® Inhaler With the Pharmacokinetics and the Safety of the Single Agents, i.e. 10 μg BI 1744 CL and 5 μg Tiotropium Bromide, Delivered Via the Respimat® Inhaler Following 21 Day-treatment Periods in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Pharmacokinetics and Safety of BI 1744 CL Plus Tiotropium Bromide in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.3
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Tiotropium Bromide

ARMS (3):
- BI 1744 CL/Tiotropium FDC (Experimental)
  Interventions: Drug: BI 1744 CL/Tiotropium FDC
- BI 1744 CL (Active Comparator)
  Interventions: Drug: BI 1744 CL
- Tiotropium (Active Comparator)
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: BI 1744 CL
  Arms: BI 1744 CL
Drug: BI 1744 CL/Tiotropium FDC
  Arms: BI 1744 CL/Tiotropium FDC
Drug: Tiotropium
  Arms: Tiotropium

SUMMARY:
The purpose of this study is to compare the systemic exposure to BI 1744 BS and tiotropium at steady state following inhalation of the fixed dose combination (FDC) of 10 μg BI 1744 CL plus 5 μg tiotropium bromide with the systemic exposure to BI 1744 BS and tiotropium at steady state following inhalation of the single agents, i.e., 10 μg BI 1744 CL and 5 μg tiotropium bromide, when administered once-daily via the Respimat® Inhaler for 21 days.

The secondary objectives were to compare the safety and tolerability (adverse events, 12-lead electrocardiogram recordings, pulmonary function testing) of BI 1744 CL and tiotropium bromide when administered as fixed dose combination or as single-agent therapy.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with International Conference on Harmonisation (ICH) - Good Clinical Practice (GCP) guidelines and local legislations prior to any study-related procedures, which includes medication washout and restrictions
2. All patients must have a diagnosis of COPD and must meet the following spirometric criteria: Patients must have relatively stable airway obstruction with a post-bronchodilator forced expiratory volume in one second (FEV1) ≥ 30 % of predicted normal and < 80% of predicted normal and a post-bronchodilator FEV1 / forced vital capacity (FVC) < 70% at Visit 1
3. Male or female patients, 40 years of age or older
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack years
5. Patients must be able to perform technically acceptable pulmonary function tests during the study period as required in the protocol
6. Patients must be able to inhale medication in a competent manner from the Respimat® inhaler and from a metered dose inhalator (MDI)

Exclusion Criteria:

1. Patients with a significant disease other than COPD; a significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the study, (ii) influence the results of the study, or (iii) cause concern regarding the patient's ability to participate in the study
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry or urinalysis; all patients with a serum glutamic oxaloacetic transaminase (SGOT) > 2.5 x ULN, serum glutamic pyruvic transaminase (SGPT) > 2.5 x ULN, bilirubin >2x upper limit of normal (ULN), creatinine >2 x ULN or creatinine clearance < 50 mL/min (Estimation of Glomerular Filtration Rate (GFR) by using the Cockcroft-Gault Formula) will be excluded regardless of clinical condition (a repeat laboratory evaluation will not be conducted in these patients)
3. Patients with a history of asthma or a total blood eosinophil count ≥600/mm3
4. Patients with any of the following conditions:

   * a diagnosis of thyrotoxicosis
   * a diagnosis of paroxysmal tachycardia (>100 beats per minute)
   * a marked baseline prolongation of QT/QTc interval
   * a history of additional risk factors for Torsade de Pointes (TdP) (e.g. heart failure, hypokalaemia, family history of Long QT Syndrome)
5. Patients with any of the following conditions:

   * a history of myocardial infarction within 1 year of screening visit (Visit 1)
   * a diagnosis of cardiac arrhythmia, arterial hypertension or coronary heart disease
   * known active tuberculosis
   * a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed)
   * a history of life-threatening pulmonary obstruction
   * a history of cystic fibrosis
   * clinically evident bronchiectasis
   * a history of significant alcohol or drug abuse
6. Patients who have undergone thoracotomy with pulmonary resection
7. Patients being treated with any of the following concomitant medications:

   * medications that prolong the QT/QTc interval since the effects of BI 1744 CL on QT/QTc interval have yet to be fully characterized
   * oral β-adrenergics
   * β-blockers (topical β -blockers for ocular conditions are allowed)
   * oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
8. Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits
9. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the Screening Visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program
10. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit (Visit 1)
11. Patients with known hypersensitivity to β-adrenergics and/or anticholinergic drugs, benzalkonium chloride, ethylenediaminetetraacetic acid or any other component of the Respimat® inhalation solution delivery system
12. Pregnant or nursing women
13. Women of childbearing potential not using two highly effective methods of birth control (one barrier and one non-barrier). Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomised partner. Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years
14. Patients who have previously been randomized in this study or are currently participating in another study
15. Patients who are unable to comply with pulmonary medication restrictions prior to randomization
16. According to Inclusion Criterion No. 2, patients with a post-bronchodilator FEV1 of < 30% of predicted normal will always be excluded. Patients with a post-bronchodilator FEV1 between 30 and 50% of predicted normal will be excluded from the study, if they display additional symptoms of chronic respiratory insufficiency or right ventricular insufficiency
17. Patients with narrow angle glaucoma, prostate hyperplasia, or bladder neck obstruction

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A randomised, double-blind, 3-way crossover study, each patient received each of the three treatments for 21 days according to randomisation.
Groups:
- Tio+Olo 5/10 μg, Olo 10 μg, Tio 5 μg: Patients received a total of three treatments, the treatments which were administered by oral inhalation, from the Respimat inhaler once daily, in the morning for 21 days, were:
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 10 µg
  * Olodaterol (Olo) 10 µg.
  * Tiotropium (Tio) 5 µg.
- Tio+Olo 5/10 μg, Tio 5 μg, Olo 10 μg: Patients received a total of three treatments, the treatments which were administered by oral inhalation, from the Respimat inhaler once daily, in the morning for 21 days, were:
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 10 µg
  * Tiotropium 5 µg.
  * Olodaterol 10 µg.
- Olo 10 μg, Tio+Olo 5/10 μg, Tio 5 μg: Patients received a total of three treatments, the treatments which were administered by oral inhalation, from the Respimat inhaler once daily, in the morning for 21 days, were:
  * Olodaterol 10 µg.
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 10 µg
  * Tiotropium 5 µg.
- Olo 10 μg, Tio 5 μg, Tio+Olo 5/10 μg: Patients received a total of three treatments, the treatments which were administered by oral inhalation, from the Respimat inhaler once daily, in the morning for 21 days, were:
  * Olodaterol 10 µg.
  * Tiotropium 5 µg.
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 10 µg
- Tio 5 μg, Tio+Olo 5/10 μg, Olo 10 μg: Patients received a total of three treatments, the treatments which were administered by oral inhalation, from the Respimat inhaler once daily, in the morning for 21 days, were:
  * Tiotropium 5 µg.
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 10 µg
  * Olodaterol 10 µg.
- Tio 5 μg, Olo 10 μg, Tio+Olo 5/10 μg: Patients received a total of three treatments, the treatments which were administered by oral inhalation, from the Respimat inhaler once daily, in the morning for 21 days, were:
  * Tiotropium 5 µg.
  * Olodaterol 10 µg.
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 10 µg
Period: Treatment Period 1 (21 Days)
Arm/Group | Tio+Olo 5/10 μg, Olo 10 μg, Tio 5 μg | Tio+Olo 5/10 μg, Tio 5 μg, Olo 10 μg | Olo 10 μg, Tio+Olo 5/10 μg, Tio 5 μg | Olo 10 μg, Tio 5 μg, Tio+Olo 5/10 μg | Tio 5 μg, Tio+Olo 5/10 μg, Olo 10 μg | Tio 5 μg, Olo 10 μg, Tio+Olo 5/10 μg
Started | 8 | 7 | 8 | 7 | 8 | 9
Completed | 8 | 7 | 8 | 7 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (21 Days)
Arm/Group | Tio+Olo 5/10 μg, Olo 10 μg, Tio 5 μg | Tio+Olo 5/10 μg, Tio 5 μg, Olo 10 μg | Olo 10 μg, Tio+Olo 5/10 μg, Tio 5 μg | Olo 10 μg, Tio 5 μg, Tio+Olo 5/10 μg | Tio 5 μg, Tio+Olo 5/10 μg, Olo 10 μg | Tio 5 μg, Olo 10 μg, Tio+Olo 5/10 μg
Started | 8 | 7 | 8 | 7 | 8 | 9
Completed | 8 | 7 | 8 | 7 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (21 Days)
Arm/Group | Tio+Olo 5/10 μg, Olo 10 μg, Tio 5 μg | Tio+Olo 5/10 μg, Tio 5 μg, Olo 10 μg | Olo 10 μg, Tio+Olo 5/10 μg, Tio 5 μg | Olo 10 μg, Tio 5 μg, Tio+Olo 5/10 μg | Tio 5 μg, Tio+Olo 5/10 μg, Olo 10 μg | Tio 5 μg, Olo 10 μg, Tio+Olo 5/10 μg
Started | 8 | 7 | 8 | 7 | 8 | 9
Completed | 8 | 7 | 8 | 7 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set. All randomised patients who received at least one dose of trial medication were included in the treated set.
Groups:
- All Subjects: A randomised, active-controlled, double-blind, 3-way crossover study in patients with COPD (chronic obstructive pulmonary disease). All participants received each of the three treatment arms in a randomly assigned order, the three treatments, which were administered by oral inhalation, from the Respimat inhaler once daily, in the morning for 21 days, were:
  * Fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 10 µg
  * Olodaterol 10 µg.
  * Tiotropium 5 µg.
Arm/Group | All Subjects
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-1h,ss) of Olodaterol
Description: Area under the concentration time curve of Olodaterol in plasma over the time interval t1=0 to t2=1 hour at steady state (AUC(0-1h,ss)).
  As plasma concentrations were not expected to be quantifiable over the complete dosing interval in all patients, t2 was defined as the time-point where at least 2/3 of the patients reveal quantifiable plasma concentrations of Olodaterol. Based on the given definition AUC(0-1h,ss) was selected as primary endpoint.
  The displayed values show adjusted gMeans and intra-subject variabilities calculated from the statistical model (ANOVA).
Time Frame: Within 30 min before drug administration and 0:02, 0:05, 0:10, 0:15, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00 hours after drug administration on Day 21 of the actual treatment period.
Population: Pharmacokinetic (PK) set which included all patients in the treated set who provided at least one of the PK parameters in at least one treatment period and completed the trial without any important protocol violations, it is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Groups:
- Tiotropium+Olodaterol 5/10 μg: Oral inhalation of fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 10 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning, for 21 days.
- Olodaterol 10 µg: Oral inhalation of Olodaterol 10 µg (5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning, for 21 days.
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg
Number analyzed (Participants) | 39 | 37
pg*h/mL | 4.67 (32.15) | 4.15 (32.15)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol 5/10 μg vs Olodaterol 10 µg; Comparison of Olodaterol (Tiotropium+Olodaterol 5/10 μg: Olodaterol 10 µg). No formal testing; Test type: Superiority or Other; ANOVA; ANOVA on the logarithmic scale with fixed effect for treatment, period, sequence, centre and random effect for subject within sequence and centre; Geometric Mean Ratio = 1.12, 90% CI 2-sided [0.99 to 1.27], Standard Deviation 32.15 — The standard deviation is actually the geometric intra-individual coefficient of variation

2. Primary Outcome: Cmax,ss of Olodaterol
Description: Maximum measured concentration of Olodaterol in plasma at steady state (Cmax,ss).
  The displayed values show adjusted gMeans and intra-subject variabilities calculated from the statistical model (ANOVA).
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg
Number analyzed (Participants) | 45 | 44
pg/mL | 5.87 (27.17) | 5.28 (27.17)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol 5/10 μg vs Olodaterol 10 µg; Comparison of Olodaterol (Tiotropium+Olodaterol 5/10 μg: Olodaterol 10 µg). No formal testing; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 1.11, 90% CI 2-sided [1.01 to 1.22], Standard Deviation 27.17 — The standard deviation is actually the geometric intra-individual coefficient of variation

3. Primary Outcome: Ae(0-24h,ss) of Tiotropium
Description: Amount of Tiotropium that was eliminated in urine at steady state from time point 0 to 24 h post-inhalation (Ae(0-24h,ss)).
  The displayed values show adjusted gMeans and intra-subject variabilities calculated from the statistical model (ANOVA).
Time Frame: Intervals 0-4, 4-8, 8-12 and 12-24 hours on Day 21 of the actual treatment period.
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Groups:
- Tiotropium 5 µg: Oral inhalation of Tiotropium 5 µg (2.5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning, for 21 days.
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Tiotropium 5 µg
Number analyzed (Participants) | 45 | 43
ng | 900.57 (20.43) | 918.63 (20.43)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol 5/10 μg vs Tiotropium 5 µg; Comparison of Tiotropium (Tiotropium+Olodaterol 5/10 μg: Tiotropium 5 µg). No formal testing; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.98, 90% CI 2-sided [0.91 to 1.06], Standard Deviation 20.43 — The standard deviation is actually the geometric intra-individual coefficient of variation

4. Secondary Outcome: Ae(0-24h,ss) of Olodaterol
Description: Amount of Olodaterol that was eliminated in urine at steady state from time point 0 to 24 h post-inhalation (Ae(0-24h,ss)).
  The displayed values show adjusted gMeans and intra-subject variabilities calculated from the statistical model (ANOVA).
Time Frame: Intervals 0-4, 4-8, 8-12 and 12-24 hours on Day 21 of the actual treatment period.
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg
Number analyzed (Participants) | 46 | 43
ng | 360.98 (19.85) | 344.17 (19.85)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol 5/10 μg vs Olodaterol 10 µg; Comparison of Olodaterol (Tiotropium+Olodaterol 5/10 μg: Olodaterol 10 µg). No formal testing; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 1.05, 90% CI 2-sided [0.98 to 1.13], Standard Deviation 19.85 — The standard deviation is actually the geometric intra-individual coefficient of variation

5. Secondary Outcome: AUC(0-6h,ss) of Tiotropium
Description: Area under the concentration time curve of Tiotropium in plasma over the time interval t1=0 to t2=6 h at steady state (AUC(0-6h,ss)).
  As plasma concentrations were not expected to be quantifiable over the complete dosing interval in all patients, t2 was defined as the time-point where at least 2/3 of the patients reveal quantifiable plasma concentrations of Tiotropium. Based on the given definition AUC(0-6h,ss) was selected as secondary endpoint.
  The displayed values show adjusted gMeans and intra-subject variabilities calculated from the statistical model (ANOVA).
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Tiotropium 5 µg
Number analyzed (Participants) | 36 | 35
pg*h/mL | 29.97 (19.81) | 33.24 (19.81)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol 5/10 μg vs Tiotropium 5 µg; Comparison of Tiotropium (Tiotropium+Olodaterol 5/10 μg: Tiotropium 5 µg). No formal testing; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.90, 90% CI 2-sided [0.83 to 0.98], Standard Deviation 19.81 — The standard deviation is actually the geometric intra-individual coefficient of variation

6. Secondary Outcome: Cmax,ss of Tiotropium
Description: Maximum measured concentration of Tiotropium in plasma at steady state (Cmax,ss).
  The displayed values show adjusted gMeans and intra-subject variabilities calculated from the statistical model (ANOVA).
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Tiotropium 5 µg
Number analyzed (Participants) | 47 | 45
pg/mL | 15.55 (29.92) | 16.15 (29.92)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol 5/10 μg vs Tiotropium 5 µg; Comparison of Tiotropium (Tiotropium+Olodaterol 5/10 μg : Tiotropium 5 µg). No formal testing; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.96, 90% CI 2-sided [0.87 to 1.07], Standard Deviation 29.92 — The standard deviation is actually the geometric intra-individual coefficient of variation

7. Secondary Outcome: AUC(0-2h,ss) of Olodaterol
Description: Area under the concentration time curve of Olodaterol in plasma over the time interval 0 to 2 hours at steady state (AUC(0-2h,ss)).
  The displayed values show adjusted gMeans and intra-subject variabilities calculated from the statistical model (ANOVA).
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg
Number analyzed (Participants) | 37 | 30
pg*h/mL | 8.52 (21.33) | 8.36 (21.33)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol 5/10 μg vs Olodaterol 10 µg; Comparison of Olodaterol (Tiotropium+Olodaterol 5/10 μg : Olodaterol 10 µg). No formal testing; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 1.02, 90% CI 2-sided [0.93 to 1.12], Standard Deviation 21.33 — The standard deviation is actually the geometric intra-individual coefficient of variation

8. Secondary Outcome: AUC(0-4h,ss) of Tiotropium
Description: Area under the concentration time curve of Tiotropium in plasma over the time interval t1=0 to t2=4 h at steady state (AUC(0-4h,ss)).
  The displayed values show adjusted gMeans and intra-subject variabilities calculated from the statistical model (ANOVA).
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Tiotropium 5 µg
Number analyzed (Participants) | 44 | 39
pg*h/mL | 21.92 (22.61) | 24.00 (22.61)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol 5/10 μg vs Tiotropium 5 µg; Comparison of Tiotropium (Tiotropium+Olodaterol 5/10 μg : Tiotropium 5 µg). No formal testing; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.91, 90% CI 2-sided [0.84 to 1.00], Standard Deviation 22.61 — The standard deviation is actually the geometric intra-individual coefficient of variation

9. Secondary Outcome: AUC(0-tz,ss) of Olodaterol
Description: Area under the plasma concentration-time curve at steady state over the time interval from 0 to the time of the last quantifiable data point (AUC(0-tz)) for Olodaterol.
  The displayed values show adjusted gMeans and intra-subject variabilities calculated from the statistical model (ANOVA).
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg
Number analyzed (Participants) | 45 | 44
pg*h/mL | 12.20 (96.12) | 9.25 (96.12)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol 5/10 μg vs Olodaterol 10 µg; Comparison of Olodaterol (Tiotropium+Olodaterol 5/10 μg; Olodaterol 10 µg). No formal testing; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio = 1.32, 90% CI 2-sided [0.98 to 1.77], Standard Deviation 96.12 — The standard deviation is actually the geometric intra-individual coefficient of variation

10. Secondary Outcome: AUC(0-tz,ss) of Tiotropium
Description: Area under the plasma concentration-time curve at steady state over the time interval from 0 to the time of the last quantifiable data point (AUC(0-tz)) for Tiotropium.
  The displayed values show adjusted gMeans and intra-subject variabilities calculated from the statistical model (ANOVA).
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Tiotropium 5 µg
Number analyzed (Participants) | 47 | 45
pg*h/mL | 32.67 (72.08) | 32.91 (72.08)
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol 5/10 μg vs Tiotropium 5 µg; Comparison of Tiotropium (Tiotropium+Olodaterol 5/10 μg; Tiotropium 5 µg). No formal testing; Test type: Superiority or Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.99, 90% CI 2-sided [0.79 to 1.24], Standard Deviation 72.08 — The standard deviation is actually the geometric intra-individual coefficient of variation

11. Secondary Outcome: Tmax,ss of Olodaterol
Description: Time from dosing to the maximum concentration of Olodaterol in plasma at steady state (tmax,ss).
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Median (Full Range); unit: h
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg
Number analyzed (Participants) | 45 | 44
h | 0.25 [0.050 to 2.020] | 0.25 [0.083 to 1.000]

12. Secondary Outcome: Tmax,ss of Tiotropium
Description: Time from dosing to the maximum concentration of Tiotropium in plasma at steady state (tmax,ss).
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Median (Full Range); unit: h
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Tiotropium 5 µg
Number analyzed (Participants) | 47 | 45
h | 0.083 [0.033 to 0.333] | 0.083 [0.033 to 0.333]

13. Secondary Outcome: fe(0-24,ss) of Olodaterol
Description: Fraction of Olodaterol eliminated in urine from 0 to 24 hours at steady state (fe(0-24,ss)).
  The displayed values show gMeans and inter-subject variabilities calculated from descriptive statistics.
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of olodaterol dose
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg
Number analyzed (Participants) | 46 | 43
percentage of olodaterol dose | 3.62 (43.8) | 3.57 (47.7)

14. Secondary Outcome: fe(0-24,ss) of Tiotropium
Description: Fraction of Tiotropium eliminated in urine from 0 to 24 hours at steady state (fe(0-24,ss)).
  The displayed values show gMeans and inter-subject variabilities calculated from descriptive statistics.
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of tiotropium dose
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Tiotropium 5 µg
Number analyzed (Participants) | 45 | 43
percentage of tiotropium dose | 18.2 (41.5) | 18.6 (46.1)

15. Secondary Outcome: Cmin,ss of Olodaterol
Description: Minimum concentration of the analyte in plasma at steady state over a uniform dosing interval (Cmin,ss).
  The displayed values show gMeans and inter-subject variabilities calculated from descriptive statistics.
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg
Number analyzed (Participants) | 45 | 44
pg/mL | 2.30 (12.6) | 2.26 (12.0)

16. Secondary Outcome: Cmin,ss of Tiotropium
Description: as for outcome 15
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Tiotropium 5 µg
Number analyzed (Participants) | 47 | 45
pg/mL | 2.95 (14.9) | 2.89 (9.84)

17. Secondary Outcome: Tmin,ss of Olodaterol
Description: Time from last dosing to the minimum concentration of the analyte in plasma at steady state over a uniform dosing interval (tmin,ss)
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Median (Full Range); unit: h
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg
Number analyzed (Participants) | 45 | 44
h | 2.00 [0.0 to 24.0] | 1.01 [0.0 to 12.0]

18. Secondary Outcome: Tmin,ss of Tiotropium
Description: as for outcome 17
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Median (Full Range); unit: h
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Tiotropium 5 µg
Number analyzed (Participants) | 47 | 45
h | 6.00 [0.0 to 24.0] | 8.00 [0.33 to 24.0]

19. Secondary Outcome: Concentration of Olodaterol in Plasma
Description: Concentration of the analyte in plasma at 0.333 hours (20 minutes) after the 8th, 14th and 21st dose, C(0.333_8), C(0.333_14,ss) and C(0.333_21,ss) respectively. As steady state was anticipated to be reached by day 14 at the latest, the index 'ss' was used for days 14 and 21.
  The displayed values show gMeans and inter-subject variabilities calculated from descriptive statistics.
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg
Number analyzed (Participants) | 43 | 40
pg/mL
  C(0.333_8) (N=38, 34) | 5.09 (48.0) | 4.48 (48.2)
  C(0.333_14,ss) (N=41, 38) | 5.13 (41.4) | 4.66 (52.5)
  C(0.333_21,ss) (N=43, 40) | 5.23 (53.7) | 4.80 (54.5)

20. Secondary Outcome: Concentration of Tiotropium in Plasma
Description: as for outcome 19
Time Frame: as for outcome 1
Population: Pharmacokinetic set which is however restricted to patients with evaluable data for this endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Tiotropium 5 µg
Number analyzed (Participants) | 46 | 44
pg/mL
  C(0.333_8) (N=40, 38) | 8.90 (60.7) | 9.58 (52.9)
  C(0.333_14,ss) (N=43, 40) | 9.08 (53.3) | 9.02 (60.3)
  C(0.333_21,ss) (N=46, 44) | 8.34 (53.2) | 9.21 (58.8)

21. Secondary Outcome: FVC Change From Baseline
Description: Mean change from baseline in forced vital capacity (FVC). Pulmonary function test.
  The baseline value was measured pre-dose on day 1 of the first treatment period.
Time Frame: 0:30 and 1:00 h after drug administration on the first day of each treatment period
Population: Treated Set.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg | Tiotropium 5 µg
Number analyzed (Participants) | 47 | 47 | 47
L
  0:30 h after drug administration (N=47, 47, 47) | 0.485 (0.354) | 0.450 (0.406) | 0.436 (0.321)
  1:00 h after drug administration (N=47, 46, 47) | 0.547 (0.409) | 0.522 (0.375) | 0.470 (0.387)

22. Secondary Outcome: FEV1 Change From Baseline
Description: Mean change from baseline in forced expiratory volume in one second (FEV1). Pulmonary function test.
  The baseline value was measured pre-dose on day 1 of the first treatment period.
Time Frame: 0:30 and 1:00 h after drug administration on the first day of each treatment period
Population: Treated Set.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg | Tiotropium 5 µg
Number analyzed (Participants) | 47 | 47 | 47
L
  0:30 h after drug administration (N=47, 47, 47) | 0.275 (0.202) | 0.292 (0.233) | 0.271 (0.211)
  1:00 h after drug administration (N=47, 46, 47) | 0.335 (0.250) | 0.357 (0.237) | 0.284 (0.206)

23. Secondary Outcome: Clinical Relevant Abnormalities in Vital Signs, Physical Examination, Blood Chemistry, Haematology, Urinanalysis and ECG
Description: Clinically relevant abnormalities in vital signs (blood pressure and pulse rate), physical examination, blood chemistry, haematology, urinanalysis and ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events. Any adverse events which occurred within 14 days following the last drug administration were assigned to the last study treatment administered.
Time Frame: From drug administration until 14 days following the last drug administration
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg | Tiotropium 5 µg
Number analyzed (Participants) | 47 | 47 | 47
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From drug administration until 14 days following the last drug administration were assigned to the last study treatment administered, upto 37 days.
Description: At each visit, all adverse events, regardless of causality, were recorded on the adverse event case report form page after discussion with the patient.
Arm/Group | Tiotropium+Olodaterol 5/10 μg | Olodaterol 10 µg | Tiotropium 5 µg
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 6/47 | 10/47 | 9/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium+Olodaterol 5/10 μg (N=47) | Olodaterol 10 µg (N=47) | Tiotropium 5 µg (N=47)
Nasopharyngitis (Infections and infestations) | 2 | 4 | 3
Headache (Nervous system disorders) | 3 | 3 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1

LIMITATIONS AND CAVEATS:
Additional secondary endpoints were listed in the original protocol, but according to internal rules, descriptive statistics would not be calculated unless data from at least 2/3rds of all subjects were available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.